CLINICAL TRIAL: NCT00525265
Title: A Clinical Pharmacological Study of OPC-41061 in the Treatment of Cardiac Edema (Congestive Heart Failure)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-06-004
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Cardiac Edema
Keywords: Vasopressin antagonist; Cardiac Edema; Diuretics
MeSH Terms: conditions — Edema, Cardiac | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): OPC-41061
  Interventions: Drug: OPC-41061(Tolvaptan)
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-41061(Tolvaptan) — Subjects will be orally administered OPC-41061 7.5 mg or 15 mg once daily after breakfast for seven days.
  Arms: 1
Drug: Placebo — Subjects will be orally administered placebo once daily after breakfast for seven days.
  Arms: 2

SUMMARY:
To investigate the pharmacokinetics, pharmacodynamics (urine volume and fluid intake), efficacy(body weight, pulmonary congestion and other congestions including cardiothoracic ratio) and safety of 7-day repeated oral administration of OPC-41061 at 7.5 mg or 15 mg in congestive heart failure (cardiac edema) patients with extracellular volume expansion despite the use of a diuretic.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with cardiac edema receiving diuretic treatments 7 days prior to the start of treatment.
2. Subjects able to receive a daily regular dosage of furosemide at 40-mg to 80-mg from the observation period until the end-of-treatment examination.
3. CHF patients with lower limb edema, jugular venous distention, or pulmonary congestion due to extracellular volume expansion.
4. Male or female subjects between the age of 20 and 85, inclusive.
5. Subjects able to stay at the study site from the day before the start of the run-in observation period until completion of post-dosing examination 2.
6. Subjects capable of giving informed consent to participate in the study of their own free will.

Exclusion Criteria:

1. Subjects with heart failure with markedly fluctuating symptoms.
2. Subjects with an assisted circulation device.
3. Subjects with any of the following complications or symptoms:(1)Suspected decrease in circulatory blood flow,(2)Hypertrophic cardiomyopathy (other than dilated phase),(3)Cardiac valve disease with significant heart valve stenosis,(4)Hepatic coma.
4. Subjects who develop acute myocardial infarction within 30 days prior to the screening examination.
5. Subjects with well-defined diagnosis of active myocarditis or amyloid cardiomyopathy.
6. Subjects with any of the following complications or symptoms:(1)Diabetes mellitus with poorly controlled blood glucose,(2)Anuria,(3)Urination impaired due to urinary tract stricture,urinary calculus,tumor in urinary tract,or other cause.
7. Subjects with a history of any of the following diseases:(1)Sustained ventricular tachycardia or ventricular fibrillation within 30 days prior to the screening examination in patients without an implanted defibrillator,(2)Cerebrovascular disorder within 6 months prior to the screening examination (other than asymptomatic cerebral infarction),(3)Hypersensitivity or idiosyncratic reaction to benzazepine derivatives.
8. Subjects who are morbidly obese (body mass index exceeding 35).
9. Subjects with systolic blood pressure in the decubitus position below 90 mmHg.
10. Subjects with any of the following abnormal laboratory values:(1)Total bilirubin > 3.0 mg/dL,(2) serum creatinine > 3.0 mg/dL,(3)serum sodium > 147 mEq/L,(4)serum potassium > 5.5 mEq/L.
11. Subjects who are unable to take oral medication.
12. Female subjects who are pregnant, possibly pregnant, or lactating, or who plan to become pregnant.
13. Subjects who received any investigational drug other than OPC-41061 within 30 days prior to the screening examination.
14. Subjects who previously participated in this or any other study of OPC-41061 and received OPC-41061.
15. Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (2):
- Japan (2):
  - Kanto Region
  - Kyushu Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-41061 7.5 mg: OPC-41061 7.5 mg/day
- OPC-41061 15 mg: OPC-41061 1.5 mg/day
Period: Overall Study
Arm/Group | OPC-41061 7.5 mg | OPC-41061 15 mg
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OPC-41061 15 mg: OPC-41061 15 mg/day
- Total: Total of all reporting groups
Arm/Group | OPC-41061 7.5 mg | OPC-41061 15 mg | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 6 | 6 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (13.6) | 66.8 (10.2) | 68.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  Japan | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: The body weight change from baseline at the time of final trial drug administration
Time Frame: Baseline, at the time of final trial drug administration
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | OPC-41061 7.5 mg | OPC-41061 15 mg
Number analyzed (Participants) | 10 | 10
Kg | -1.68 (1.83) | -2.14 (1.45)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | OPC-41061 7.5 mg | OPC-41061 15 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-41061 7.5 mg (N=10) | OPC-41061 15 mg (N=10)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-41061 7.5 mg (N=10) | OPC-41061 15 mg (N=10)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling Hot (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 1 (1)
Thirst (General disorders) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 2 (2) | 4 (5)
Blood Potassium Increased (Investigations) | 1 (1) | 1 (1)
Blood Pressure Decreased (Investigations) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 2 (2) | 5 (5)
Blood Uric Acid Increased (Investigations) | 0 (0) | 1 (1)
Blood Urine Present (Investigations) | 1 (1) | 0 (0)
Faecal Occult Blood (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Altered State of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Oedema Genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dematitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Wound Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No